CLINICAL TRIAL: NCT02595099
Title: Feasibility and Acceptability of a Mindfulness-based Intervention for People With Osteoarthritis (OA) Related Knee Pain.
Brief Title: Mindfulness for Osteoarthritis-related Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15098
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2015-05

CONDITIONS: Osteoarthritis; Chronic Pain
MeSH Terms: conditions — Osteoarthritis; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness training (Experimental): 8 week programme of Mindfulness training
  Interventions: Other: Mindfulness training

INTERVENTIONS:
Other: Mindfulness training — group-based training programme, 2.5 hours delivered weekly for 8 weeks

SUMMARY:
The purpose of this project is to investigate the feasibility and acceptability of a Mindfulness based intervention for people who are attending secondary care with Osteoarthritis (OA)-related knee pain.

DETAILED DESCRIPTION:
This study will explore the acceptability of a novel intervention (an 8-week programme of Mindfulness training) for people with Osteoarthritis(OA)-related knee pain. Mindfulness interventions provide intensive training in mindfulness meditation and its applications for coping with stress, illness and pain in day to day life. The aim of the intervention is not reduce the severity of pain per se, but to change how an individual responds and copes with pain. If effective, patients may report improvements in pain, sleep, quality of life and their ability to cope with pain in daily life.

Before carrying out a study to determine if such an intervention is effective, it is important to explore whether it is acceptable to patients. Treatments for OA knee are usually targeted at the painful joint e.g medication, injections, physiotherapy, surgery and ultimately total knee replacement (TKR), so some patients may not expect a programme based on meditation practice to help.

The investigators will recruit two groups of patients with OA-related knee pain from hospital clinics, (i) those with moderate-severe knee pain who have not yet had a TKR and (ii) those who have had a TKR who have persistent pain after one-year. All participants will complete baseline assessments before commencing an eight-week group based programme of Mindfulness training, delivered by an NHS physiotherapist who is also a trained Mindfulness teacher. Participants will have daily meditation practices to carry out at home. Follow-up questionnaires will be repeated after the intervention and again at 6 months.

After the intervention, the investigators will conduct group discussions with some of the participants to explore their expectations and experiences of the intervention and the study. Participants will be in the study for approximately 8 months (from time of recruitment) and the study will last 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years, there is no upper age limit.
* Osteoarthritis of the knee (defined as joint space narrowing and osteophytes in 1 or more compartment) and moderate to severe knee pain (defined as 40-80mm on a 100mm visual analogue scale).

Or

* Persistent moderate to severe knee pain (40 - 80mm on a 100mm visual analogue scale), one year following total knee replacement

Exclusion Criteria:

* People who have previously participated in a 8 week Mindfulness course
* Terminal illness and other conditions leading to incapacity to participate in the study
* Acute knee injury, knee joint surgery or steroid injection to the knee within previous 3 months or currently on a waiting list for knee joint surgery
* Inflammatory arthritis (eg Rheumatoid arthritis or psoriatic arthritis)
* Patients who are unable to provide informed consent
* Patients who are unable to communicate in English, as the intervention is delivered in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Acceptability | 8 weeks
  This will be determined by the number of participants who completed the intervention and from focus group discussions.

SECONDARY OUTCOMES:
WOMAC Index | 8 weeks, 6 months
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC); a 24 item self-administered health status measure widely used in assessing pain, stiffness, and function in patients with OA of the hip or knee.
Neuropathic Pain | 8 weeks, 6 months
  Pain Detect Questionnaire; a 12 item patient-based, screening questionnaire to determine the presence of neuropathic pain components validated in knee OA
self-efficacy | 8 weeks, 6 months
  The Arthritis self-efficacy scale; a 20 item questionnaire to measure self-efficacy.
Pain Attitudes | 8 weeks, 6 months
  The Survey of Pain Attitudes; a 30 item questionnaire assessing patients attitudes and beliefs about their pain.
Pain Catastrophising | 8 weeks, 6 months
  Pain catastrophizing scale for adults; a 13 item self-report measure of the degree to which people experience pain adopt exaggerated negative interpretations of the pain. and beliefs about their pain.
Anxiety and Depression | 8 weeks, 6 months
  Hospital Anxiety and Depression (HAD) scale; A 14 item, two dimension scale developed to identify depression and anxiety among physically ill patients. Validated in several patient populations.
Sleep quality | 8 weeks, 6 months
  Pittsburgh sleep quality index; a 18 item, self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval.
EQ-5D | 8 weeks, 6 months
  Euro-Qol quality of life ; a 5 item standardised instrument applicable to a wide range of health conditions and treatments for use as a measure of health outcome.
Patient generated index | 8 weeks, 6 months
  The Patient Generated Index; an individualised instrument which rates up to 5 QOL items chosen by the respondent as being important.
health service use | 8 weeks, 6 months
  Service use questionnaire; a 10 item questionnaire to measure health and social care service use including medications.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hall, Principal Investigator — University of Nottingham

REFERENCES:
- [Background] Chiesa A, Serretti A. Mindfulness-based interventions for chronic pain: a systematic review of the evidence. J Altern Complement Med. 2011 Jan;17(1):83-93. doi: 10.1089/acm.2009.0546. PMID 21265650
- [Background] Fogarty FA, Booth RJ, Gamble GD, Dalbeth N, Consedine NS. The effect of mindfulness-based stress reduction on disease activity in people with rheumatoid arthritis: a randomised controlled trial. Ann Rheum Dis. 2015 Feb;74(2):472-4. doi: 10.1136/annrheumdis-2014-205946. Epub 2014 Nov 18. No abstract available. PMID 25406303
- [Background] Zangi HA, Mowinckel P, Finset A, Eriksson LR, Hoystad TO, Lunde AK, Hagen KB. A mindfulness-based group intervention to reduce psychological distress and fatigue in patients with inflammatory rheumatic joint diseases: a randomised controlled trial. Ann Rheum Dis. 2012 Jun;71(6):911-7. doi: 10.1136/annrheumdis-2011-200351. Epub 2011 Dec 20. PMID 22186709
- [Background] Schutze R, Slater H, O'Sullivan P, Thornton J, Finlay-Jones A, Rees CS. Mindfulness-Based Functional Therapy: a preliminary open trial of an integrated model of care for people with persistent low back pain. Front Psychol. 2014 Aug 4;5:839. doi: 10.3389/fpsyg.2014.00839. eCollection 2014. PMID 25136324
- [Background] Bawa FL, Mercer SW, Atherton RJ, Clague F, Keen A, Scott NW, Bond CM. Does mindfulness improve outcomes in patients with chronic pain? Systematic review and meta-analysis. Br J Gen Pract. 2015 Jun;65(635):e387-400. doi: 10.3399/bjgp15X685297. PMID 26009534
- [Background] Sofat N, Ejindu V, Kiely P. What makes osteoarthritis painful? The evidence for local and central pain processing. Rheumatology (Oxford). 2011 Dec;50(12):2157-65. doi: 10.1093/rheumatology/ker283. Epub 2011 Sep 27. PMID 21954151
- [Background] Finan PH, Buenaver LF, Bounds SC, Hussain S, Park RJ, Haque UJ, Campbell CM, Haythornthwaite JA, Edwards RR, Smith MT. Discordance between pain and radiographic severity in knee osteoarthritis: findings from quantitative sensory testing of central sensitization. Arthritis Rheum. 2013 Feb;65(2):363-72. doi: 10.1002/art.34646. PMID 22961435
- [Background] Murphy LB, Sacks JJ, Brady TJ, Hootman JM, Chapman DP. Anxiety and depression among US adults with arthritis: prevalence and correlates. Arthritis Care Res (Hoboken). 2012 Jul;64(7):968-76. doi: 10.1002/acr.21685. PMID 22550055
- [Background] Hawker GA, Gignac MA, Badley E, Davis AM, French MR, Li Y, Perruccio AV, Power JD, Sale J, Lou W. A longitudinal study to explain the pain-depression link in older adults with osteoarthritis. Arthritis Care Res (Hoboken). 2011 Oct;63(10):1382-90. doi: 10.1002/acr.20298. Epub 2010 Jul 26. PMID 20662042
- [Background] Murphy SL, Lyden AK, Phillips K, Clauw DJ, Williams DA. Association between pain, radiographic severity, and centrally-mediated symptoms in women with knee osteoarthritis. Arthritis Care Res (Hoboken). 2011 Nov;63(11):1543-9. doi: 10.1002/acr.20583. PMID 22034116
- [Background] Wylde V, Hewlett S, Learmonth ID, Dieppe P. Persistent pain after joint replacement: prevalence, sensory qualities, and postoperative determinants. Pain. 2011 Mar;152(3):566-572. doi: 10.1016/j.pain.2010.11.023. Epub 2011 Jan 15. PMID 21239114
- [Background] Hawker G, Wright J, Coyte P, Paul J, Dittus R, Croxford R, Katz B, Bombardier C, Heck D, Freund D. Health-related quality of life after knee replacement. J Bone Joint Surg Am. 1998 Feb;80(2):163-73. doi: 10.2106/00004623-199802000-00003. PMID 9486722
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770